CLINICAL TRIAL: NCT01454726
Title: A Random Controlled Clinical Trial:l Traditional Chinese Diaoshi Jifa Therapy of Meniere's Disease
Brief Title: Clinical Trial of Traditional Chinese Diaoshi Jifa Therapy of Meniere's Disease
Acronym: TCDMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Administration of Traditional Chinese Medicine Bureau (Other Government)
Collaborators: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jianping Jia, Professor, Beijing Administration of Traditional Chinese Medicine Bureau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JJT2010-22
Record Dates: First submitted 2011-06-01; First posted 2011-10-19 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-01

CONDITIONS: Meniere's Disease
Keywords: Dizziness; Meniere's disease; Diaoshi Jifa therapy
MeSH Terms: conditions — Meniere Disease; Dizziness | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): receiving both Diaoshi Jifa therapy and the Western medical treatment.
  Interventions: Other: Diaoshi Jifa therapy plus the Western medical treatment.
- control group (Other): receiving the Western medical treatment alone.
  Interventions: Other: drug

INTERVENTIONS:
Other: Diaoshi Jifa therapy plus the Western medical treatment. — Diaoshi Jifa treatment
  Other Names: Western medical treatment: Ginkgo 20 ml qd iv, Merision 6mg tid po
  Arms: experimental group
Other: drug — the Western medical treatment alone.
  Other Names: Western medical treatment: Ginkgo 20 ml qd iv, Merision 6mg tid po
  Arms: control group

SUMMARY:
The hypothesis of this study is that DiaoShi Jifa reduces the symptoms, such as dizziness in patients with Meniere's disease.

DETAILED DESCRIPTION:
Created by Dr. Diao, DiaoShi Jifa is a well-known traditional Chinese Medicine approach to treat dizziness in patients with chronic diseases. The investigators designed this randomized clinical trial to examine whether Diaoshi Jifa significantly decreases dizziness in patients with Meniere's disease. There are 2 arms in this trial: One arm is DiaoShi Jifa plus conventional Western medical treatment, another is conventional Western medical treatment only. The dizziness handicap inventory (DHI) will be used to evaluate the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of probable Meniere's disease
2. Must be able to receive manual treatment
3. Dizziness Patients receiving other treatment longer than 5 days before entering the study.

Exclusion Criteria:

1. Patients with critical illness of internal medicine and surgery
2. Patients with spinal disease or other conditions that cannot receive manual treatment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, MD, Principal Investigator — Beijing Xuan Wu Hosipital
Locations (1):
- Xuan Wu Hosipital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: Jan 1, 2011-November 30, 2011 recruitment location: Department of Neurology, Xuan Wu Hospital of Capital Medical University
Pre-assignment Details: A total of 27 patients were enrolled and randomly attributed to either experimental or control group.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 16 | 11
Completed | 16 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 49.75 (12.63) | 54.00 (8.91) | 51.48 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  China | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Dizziness Handicap Inventory (DHI) Questionnaire Score
Description: dizziness Handicap Inventory (DHI) evaluates the self-perceived handicapping effects imposed by vestibular system disease. We employed the final version of DHI, which contains 25 items including 7 physical questions, 9 functional questions and 9 emotional questions. DHI has a total score of 100 points (4 points for each item). Higher scores indicate more severe handicap. Thus the maximum score for DHI is 100, while the minimum core is 0.
Time Frame: 0 and 24 hours
Population: Among the 27 participants enrolled in the study, one participant quitted the study before treatment application. Twenty-six patients fulfilled all the procedures and were eligible for the full analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 16 | 10
units on a scale | 10.25 (9.77) | 49.6 (20.50)

ADVERSE EVENTS:
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/10

LIMITATIONS AND CAVEATS:
Our study focused only on the effect of Diaoshi Jifa on Meniere's disease after one-time treatment. There still possibilities that after several days' treatment, both experimental and control groups have similar improvement in their DHI scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No